CLINICAL TRIAL: NCT05475314
Title: A Postbiotic Fermented Oat Gruel May Have a Beneficial Effect on the Colonic Mucosal Barrier in Patients With Irritable Bowel Syndrome
Brief Title: Effect of Postbiotic Product on Colonic Barriers in IBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nordisk Rebalance A/S (Industry)
Collaborators: University Hospital, Linkoeping (Other); Linkoeping University (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: referm-barrier
Record Dates: First submitted 2022-07-21; First posted 2022-07-26 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: IBS - Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Intervention Model Description: Patients were randomly allocated to ReFerm® (18 patients, two men) or placebo (12 patients, three men) arms. There were no significant differences between the groups in terms of age, BMI, or disease severity.
Who Masked: Participant, Care Provider
Masking Description: The appearance including colour and thickness of the two products are similar
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ReFerm(R); fermented oat gruel (Experimental): ReFerm® is manufactured by the fermentation of an oat gruel with L. plantarum 299v. The product is tested for pH and colony-forming units (CFU) of Enterobacteriaceae, yeasts/moulds, and L. plantarum 299v. The pH must be < 4.0, the CFU of Enterobacteriaceae and yeasts/moulds must be < 100/mL, and the CFU for L. plantarum 299v must be > 10E+08 immediately after completion of fermentation. The energy content of 100 mL ReFerm® is 58 kcal (240 kJ), from 1.6 g protein, 9.8 g carbohydrate, and 0.9 g fat. Each ReFerm® package contained 250 ml
  Interventions: Dietary Supplement: ReFerm(R)
- Thick-it(R); thickened water (Placebo Comparator): Thick-it ® mildly thick, Kent Precision Foods Group, Inc.; commercially available) was chosen as a placebo to mimic the viscosity. This product contains artesian mineral water and ≤ 2% xanthan gum, calcium chloride, malic acid, potassium benzoate, potassium sorbate (to preserve freshness), sodium hexametaphosphate, and disodium EDTA. The energy content of 237 mL Thick-it ® (one package) was 5 kcal (21 kJ) from 0 g protein, 1 g carbohydrate, and 0 g fat
  Interventions: Dietary Supplement: ReFerm(R)

INTERVENTIONS:
Dietary Supplement: ReFerm(R) — Enemas of approx 250 mL twice daily
  Other Names: Profermin(R)

SUMMARY:
Impaired intestinal permeability and microbial dysbiosis are important pathophysiological mechanisms underlying irritable bowel syndrome (IBS). ReFerm®, also called Profermin®, is a postbiotic product of oat gruel fermented with Lactobacillus plantarum 299v. In this experimental study, we investigated whether ReFerm® has a beneficial effect on the intestinal epithelial barrier function in patients with IBS.

DETAILED DESCRIPTION:
A single-blinded, randomised experimental study was conducted. Potential participants were screened based on the inclusion and exclusion criteria during telephone interviews. As the patients were their own controls, self-reported allergy was not an exclusion criterion as long as both interventions were carried out during unchanged allergic exposure.

Patients were then randomly allocated to one of two study arms: Referm® or thickened water (Thick-it ®, commercially available; Kent Precision Foods Group, Inc., Muscatine, IA, USA) as placebo. The patients underwent sigmoidoscopy with biopsies obtained from the distal colon at baseline and after 14 days of intervention with ReFerm® or placebo enema twice a day. The enema was administered rectally, in the left side position, and retained for as long as possible (at least 10 min) both in the left-sided and supine body position to activate retrograde peristalsis. To assess clinical improvement of symptoms, questionnaires were completed twice: before and after the intervention. During the 14 days of the intervention, the patients completed daily questionnaires. To improve compliance with the study intervention, the patients were given a check-up call by a principal investigator (OBe) twice per week during the intervention period.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed IBS-D or IBS-M according to Rome IV criteria
* Moderate to severe IBS according to IBS-SSS score (≥175p)
* Age 18-70 years
* Fluency in written and spoken Swedish language

Exclusion Criteria:

* Organic gastrointestinal disease
* Previous major gastrointestinal operation (apart from appendectomy and cholecystectomy)
* Psychiatric disease (bipolar disease, schizophrenia)
* NSAID intake less than 2 weeks prior to endoscopy
* Self-reported pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Intestinal permeability | 14 days
  Basic Science.
  Mucosal permeability change (transcellular (amount of HRP (fmol/mL) and paracellular (amount of FITC (pM)), before and after treatment using an Ussing chamber with mounted patient biopsies

SECONDARY OUTCOMES:
Symptom change | 14 days
  Symptom change using the following questionnaires systems.
  IBS severity scoring system for symptom change (significant if > 50 points) before and after treatment.
  Gastrointestinal Symptom Rating Scale-IBS and Visceral sensitivity index. Data analyzed by cluster or as a total score for all items with statistically significant change.
  Hospital Anxiety and Depression Scale. Cut-off values are indicated as ≥8 for subclinical (suspicious) anxiety or depression and ≥11 as definite cases on both the HADS-D and HADS-A, respectively.
  Short Health Scale. Data analyzed by cluster or as a total score for all items with statistically significant change.

CONTACTS AND LOCATIONS:
Overall Officials: Susanna Walter, MD, Study Chair — University Hospital, Linköping, Sweden
Locations (1):
- Linköping University Hospital, Linköping, Sweden, Linköping, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Biskou O, Walter S, Israelsen H, Winberg ME, Bednarska O, Keita AV. ReFerm(R): a postbiotic fermented oat gruel composition is reducing mast cell degranulation in the colon of patients with irritable bowel syndrome. Front Med (Lausanne). 2024 Jul 4;11:1408623. doi: 10.3389/fmed.2024.1408623. eCollection 2024. PMID 39026547
- [Derived] Bednarska O, Biskou O, Israelsen H, Winberg ME, Walter S, Keita AV. A postbiotic fermented oat gruel may have a beneficial effect on the colonic mucosal barrier in patients with irritable bowel syndrome. Front Nutr. 2022 Dec 8;9:1004084. doi: 10.3389/fnut.2022.1004084. eCollection 2022. PMID 36570171